CLINICAL TRIAL: NCT03326648
Title: The Role of Muscle Protein Breakdown in the Regulation of Muscle Quality in Frail Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truls Raastad (Other)
Collaborators: University of Padova (Other); University of Copenhagen (Other); Tine (Industry)
Responsible Party: Sponsor-Investigator, Truls Raastad, Prof., Norwegian School of Sport Sciences
Organization: Norwegian School of Sport Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STAS
Record Dates: First submitted 2017-05-05; First posted 2017-10-31 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Frailty; Strength training; Autophagy
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Subjects and testers will not be blinded. All analyses of muscle samples will be performed blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training + protein supplement (Experimental): Two sessions of strength training each week in addition to daily protein supplementation for 10 weeks.
  Interventions: Other: Strength training; Dietary Supplement: Protein supplementation
- Protein supplement (Experimental): Daily protein supplementation for 10 weeks.
  Interventions: Dietary Supplement: Protein supplementation

INTERVENTIONS:
Other: Strength training — Heavy load strength training performed twice a week for 10 weeks.
  Other Names: Resistance training
  Arms: Strength training + protein supplement
Dietary Supplement: Protein supplementation — Dietary protein supplement (protein-enriched milk with 0,2 % fat). 0,33 l each day for 10 weeks.

SUMMARY:
The purpose of this study is to investigate mechanisms underlying the reduction in muscle quality (the ratio between muscle strength and muscle size) with aging, and to investigate how these factors are affected by strength training and protein supplementation. It is already established that muscle quality defined as the ratio between the strength and the size of a muscle is improved with strength training, even in frail elderly individuals. However, the relative contribution of factors such as activation level, fat infiltration, muscle architecture and single fiber function is unknown. The main focus of this study is to investigate the relationship between muscle quality and muscle protein breakdown, as insufficient degradation of proteins is hypothesized to negatively affect muscle quality.

DETAILED DESCRIPTION:
Aging is associated with impaired skeletal muscle function. This is evident not only by a reduced capacity to generate force and power at the whole muscle level, but also by a decline in individual muscle fiber contraction velocity and force generation. Combined with muscle atrophy, these changes lead to reduced muscle strength and quality and loss off physical function with age. Clinically, muscle quality may be a better indicator of overall functional capacity than absolute muscle strength. Thus, identifying the mechanisms underlying the age-related loss of muscle quality is of high relevance for the prevention of functional impairment with aging. The explanation for the loss of muscle quality with aging seems to be multifactorial, with alterations in voluntary muscle activation, muscle architecture, fat infiltration and impaired contractile properties of single muscle fibers being likely contributors. Single fiber specific force seems to be related to myosin heavy chain (MHC) content, which is thought to reflect the number of available cross-bridges. The reduction of single fiber specific force with aging may thus be a consequence of reduced synthesis of MHC and/or increased concentration of non-contractile tissue (e.g. intramyocellular lipids).

Some studies in mice also indicate attenuated activity in some of the pathways responsible for degradation of muscle proteins with aging (especially autophagy). As a result, damaged proteins and organelles are not removed as effectively as they should, which could ultimately compromise the muscle's ability to produce force. In addition, reduced efficiency of mitophagy and lipophagy (two specific forms of autophagy), may indirectly affect single fiber specific force, through oxidative damage by reactive oxygen species (ROS) and increased levels of intramyocellular lipids, respectively. Although animal studies indicate attenuated autophagic function, exercise seems to restore the activity in this pathway. Whether this also is the case in humans is unknown. Thus, the purpose of this study is to investigate how the different factors contributing to reduced muscle quality in frail elderly individuals, with emphasis on the relationship between muscle quality and autophagy, may be counteracted by a specific strength training program targeting muscle quality and muscle mass.

In this randomized controlled trial the investigators will aim to recruit frail elderly individuals, as muscle quality is shown to be low in this population. As a consequence, the potential for improved muscle quality is expected to be large. Subjects will be randomized to two groups; one group performing strength training twice a week for 10 weeks in addition to receiving daily protein supplementation. The other group will only receive the protein supplement. Several tests will be performed before and after the intervention period, including a test day where a biopsy is obtained both at rest, and 2.5 hours following strength training + protein supplementation or protein supplementation only. This will provide information about the regulation of muscle protein breakdown in a resting state, following protein intake and following strength training in combination with protein intake. As this will be done both before and after the training period, it will also provide information on how long-term strength training affects the activity in these systems.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65
* Frail or pre-frail according to the Fried Frailty Criteria or Short Physical Performance Battery (SPPB) score <6.
* Mini Mental State Examination score > 18

Exclusion Criteria:

* Diseases or injuries contraindicating participation
* Lactose intolerance
* Allergy to milk
* Allergy towards local anesthetics (xylocain)
* Use of anticoagulants that cannot be discontinued prior to the muscle biopsy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Single fiber specific force | Change from baseline at 10 weeks
  A measure of muscle quality at the single fiber level. Biopsies obtained from m. Vastus Lateralis

SECONDARY OUTCOMES:
Lean mass | Change from baseline at 10 weeks
  Measured by a Dual-energy X-ray absorptiometry (DXA) scan
Fat mass | Change from baseline at 10 weeks
  Measured by a Dual-energy X-ray absorptiometry (DXA) scan
Bone mineral density | Change from baseline at 10 weeks
  Measured by a Dual-energy X-ray absorptiometry (DXA) scan
Muscle strength of m. quadriceps | Change from baseline at 10 weeks
  Maximal isometric and dynamic muscle strength of m. quadriceps
Muscle size of m. quadriceps | Change from baseline at 10 weeks
  Cross-sectional area of m. quadriceps measured by a Computed Tomography scan
Fat infiltration of m. quadriceps | Change from baseline at 10 weeks
  Fat infiltration of m. quadriceps measured by a Computed Tomography scan
Muscle activation | Change from baseline at 10 weeks
  Voluntary activation level during a maximal isometric knee extension using the interpolated twitch technique
Fractional Breakdown Rate | Measured over the last 14 days of the intervention period
  Measurement of fractional breakdown rate by the use of orally provided Deuterium Oxide, biopsies and blood samples
m. Vastus Lateralis thickness | Change from baseline at 10 weeks
  Measured by ultrasound
Chair stand performance | Change from baseline at 10 weeks
  Time (sec) to stand up from a chair five times
Habitual gait velocity | Change from baseline at 10 weeks
  Time (sec) to walk 6 meters at habitual gait velocity
Maximal gait velocity | Change from baseline at 10 weeks
  Time (sec) to walk 6 meters as fast as possible
Level/cellular location of Microtubule-associated protein 1A/1B-light chain 3 (LC3) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Level/cellular location of p62/Sequestosome-1 | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Level/cellular location of Lysosome-associated membrane glycoprotein 2 (LAMP2) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Level/cellular location of forkhead box O3 (FOXO3a) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Phosphorylation status and total level of ribosomal protein S6 kinase beta-1(P70S6K) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Phosphorylation status and total level of eukaryotic elongation factor 2 (eEF-2) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Phosphorylation status and total level of eukaryotic translation initiation factor 4E-binding protein 1 (4EBP-1) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Level/cellular location of muscle RING-finger protein-1 (Murf-1) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Level/cellular location of ubiquitin (Ub) | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Blood serum glucose | Change from baseline at 10 weeks
  Fasted
Blood serum insulin | Change from baseline at 10 weeks
  Fasted
Blood plasma Hemoglobin A1c (HbA1c) | Change from baseline at 10 weeks
  Fasted
Blood serum Triglycerides | Change from baseline at 10 weeks
  Fasted
Blood serum High-density lipoproteins (HDL) | Change from baseline at 10 weeks
  Fasted
Blood serum Low-density lipoproteins (LDL) | Change from baseline at 10 weeks
  Fasted
Blood serum C-reactive protein (CRP) | Change from baseline at 10 weeks
  Fasted
forkhead box protein O3 (FOXO3A) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
forkhead box protein O1 (FOXO1) mRNA mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
hepatocyte growth factor (HGF) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
insulin-like growth factor I (IGF1) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
myostatin (MSTN) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
E3 ubiquitin-protein ligase TRIM63 (TRIM63) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
p62/Sequestosome-1 mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
muscle RING-finger protein-1 (Murf-1) protein 1 (4EBP-1) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Atrogin1 mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Microtubule-associated protein 1A/1B-light chain 3 (LC3) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
BCL2/adenovirus E1B interacting protein 3 (BNIP3) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
PTEN-induced putative kinase 1 (PINK1) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
TNF receptor associated factor 6 (TRAF6) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
transcription factor EB (Tfeb) mRNA | Before and 2.5 hours after acute training session both at baseline and after 10 weeks
  Biopsies from m. Vastus Lateralis analyzed by western blot
Intramyocellular lipids | Change from baseline at 10 weeks
  Oil-Red-O staining of muscle sections. Biopsy from m. Vastus Lateralis analyzed by immunohistochemistry
Muscle fiber type distribution | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by immunohistochemistry
Muscle fiber cross-sectional area | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by immunohistochemistry
Muscle satellite cells | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by immunohistochemistry
Myonuclei | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by immunohistochemistry
Myonuclei number | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by confocal microscopy
Myonuclei location | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by confocal microscopy
Amount of mitochondria | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by confocal microscopy
Location of mitochondria | Change from baseline at 10 weeks
  Biopsy from m. Vastus Lateralis analyzed by confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, Prof., Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No